CLINICAL TRIAL: NCT04217525
Title: Duke Spine Outcome Study (DSOS)
Acronym: DSOS
Status: Suspended | Type: Observational
Why Stopped: Temporary suspension due to staffing
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00101198
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-05

CONDITIONS: Spinal Tumor; Spinal Disorder
MeSH Terms: conditions — Spinal Cord Neoplasms; Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Will collect up to 60mL of blood and 5mL of bone marrow.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Disorders: This group includes patients with any spinal deformity or disorder coming in for treatment.
- Spinal Tumors: This group includes patients with spinal tumors or metastasis of the spine, coming in for treatment.

SUMMARY:
The primary goal of this registry is to increase the knowledge about spine tumors and other spine disorders to guide appropriate management strategies for the future. This registry will include the review of medical records, data collection for health related quality of life questionnaires, and collected tissues and samples.

The study will require obtaining spinal lesions (tumor, etc.), blood, and bone marrow samples (from non-lesional bone) from selected patients, which will be collected during your surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years.
* Able to read and write local language at an elementary level.
* Diagnosis of primary or metastatic tumor of the spine ); or
* Infection of the spine; or
* Instability of the spine; or
* Injury of the spine.
* Accessibility for treatment and follow up.
* Patient consent obtained according to Duke institutional policy.

Inclusion criteria for spine surgery (control population for bone marrow specimens)

* Age between 18 and 85 years.
* Spine surgery to be performed at Duke University Medical Center (DUMC) under the auspices of the neurosurgery program.
* No concurrent cancer diagnosis.
* Accessibility for treatment and follow up.
* Patient consent obtained according to Duke institutional policy.

Exclusion Criteria:

* History of substance abuse (recreational drugs, alcohol) within 12 months prior to screening
* Is a prisoner.
* A disease or condition that would, in opinion of the investigator, preclude accurate evaluation

  (e.g. significant psychiatric disease), or that would impair the ability of the patient to receive protocol treatment or comply with protocol.
* Pregnant or breast feeding during the study period (women of child-bearing potential will require a negative serum pregnancy test within 30 days of enrollment).
* Active infection, or fever of unknown origin.
* Inflammatory bowel disease.
* Systemic lupus erythematosus.
* Rheumatoid arthritis, or other autoimmune disease.
* History of or active hematologic or bone marrow diseases, including but not limited to diagnosed lymphomas, leukemias, sickle cell or other anemias not associated with their current condition.
* Polycythemia vera.
* Known or suspected immunodeficiency or Human Immunodeficiency Virus (HIV).
* Hematocrit < 24% pre-operatively.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spinal disorders or spinal tumors.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-12-03 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life as measured by Spine Cancer Outcomes Questionnaire (SCOQ) | Baseline, 6, 12, 26, 52, 104 weeks
  It is made up of 5 domains: physical function, neural function, pain, mental health and social function. It was developed as a comparison to the 36-Item Short Form Survey (SF-36) for patients with spine tumors. The reliability and validity of this questionnaire will be compared with the SF-36v2.
Change in Pain Score as measured by Pain Numeric Rating Scale (NRS) | Baseline, 6, 12, 26, 52, 104 weeks
  The Pain NRS is an 11-point horizontal scale where the end points are the extremes of no pain (0) and pain as bad as it could be, or worst pain (10). It measures subjective intensity of pain and the patient rates his/her overall or average daily pain.
Change in Quality of Life as measured by SF-36 version 2 | Baseline, 6, 12, 26, 52, 104 weeks
  Short-form health survey with 36 questions
Change in Health Status as measured by EQ-5D | Baseline, 6, 12, 26, 52, 104 weeks
  It contains 5 questions and provides a simple descriptive profile and a single index value for health status.
Change in Daily Living Abilities as measured by Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline, 6, 12, 26, 52, 104 weeks
  Grade 0 = Fully active to 5 = Dead
Change in Neurological Function as measured by International Standards Neurological Classification of Spinal Cord Injury (ISNCSCI) | Baseline, 6, 12, 26, 52, 104 weeks
  ISNCSCI is a standardized examination to determine neurologic function and has been a standard clinical assessment for patients with neurological deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Courtney R. Goodwin, M.D., PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No